CLINICAL TRIAL: NCT06158893
Title: Comparison of Preoperative Inhaled Budesonide With Salbutamol on the Respiratory Adverse Effects in Children Undergoing Tonsillectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ziad Shaban Redwan Helal, Resident Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: children undergo Tonsillectomy
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Preoperative Inhalation of Budesonide and Salbutamol in Children Undergoing Tonsillectomy
MeSH Terms: interventions — Albuterol; Budesonide; Sodium Chloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- salbutamol (Experimental): children will receive 0.15 milligram per kilogram of salbutamol diluted with normal saline to a total volume of 4 ml by inhalation 20 minutes preoperatively
  Interventions: Drug: Salbutamol
- budesonide (Active Comparator): children will receive 0.5 milligram per kilogram of budesonide diluted with normal saline to a total volume of 4 ml by inhalation 20 minutes preoperatively
  Interventions: Drug: Budesonide
- normal saline (Placebo Comparator): children will receive 0.4 ml of normal saline 0.9 by inhalation 20 minutes preoperatively
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Salbutamol — inhalation anaesthesia
  Arms: salbutamol
Drug: Budesonide — inhalation anaesthesia
  Arms: budesonide
Other: Saline — saline
  Arms: normal saline

SUMMARY:
Comparison of preoperative inhaled Budesonide with Salbutamol on the incidence of respiratory adverse effects in children undergoing tonsillectomy

DETAILED DESCRIPTION:
Comparison of preoperative inhaled Budesonide with Salbutamol on the incidence of respiratory adverse effects in children undergoing tonsillectomy Adenotosillectomy is routinely performed for children with sleep disordered breathing or recurrent infectious tonsillitis. Although the safety of the pediatric anesthesia is constantly improving, a substantial proportion of children undergoing tonsillectomies experience pre operative respiratory adverse events with a prevalence up to 50% in children with at least one risk factor. Both minor adverse effects such as oxygen desaturation airway, obstruction coughing or wheezing and the major events such as laryngospasm and/ or bronchospasm occur more commonly undergoing tonsillectomy compared with other non airway surgery.

ELIGIBILITY:
Inclusion Criteria:

1. children scheduled for elective tonsillectomy with or without adenoidectomy, grommets cautery of inferior turbinates.
2. Age more than or equal 5 years and less than or equal to 12 years.
3. Both genders
4. No obvious abnormalities in preoperative ECG, blood routine electrolytes and other tests.
5. ASA class 1

Exclusion Criteria:

1. Patients with Known hypersensitivity to any of the drugs that would be used in the study
2. Patients that are immunologically compromised
3. Sleep apnea syndrome or difficult airway
4. Pre-existing hypoxemia is SpO2 < 90%
5. History of adverse events with prior sedation or patients who had taken any sedative drugs within the last 24 hours.
6. Parents refusal

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
incidence of preoperative respiratory adverse events. | 1 year
  Will be the incidence of preoperative respiratory adverse events. events will be reported by the attending an anesthetist or PACU nurse on a dedicated data collection sheet and will be recorded against the phase of anesthesia (induction, maintenance, emergency, or recovery) during which the event occurred

SECONDARY OUTCOMES:
frequency of the individual PRAEs | 1 year
  Will be the frequency of the individual PRAEs, incidence of PRAEs during the induction and recovery periods, recovery time (the time from the end of surgery to discharge from PACU)